CLINICAL TRIAL: NCT06050863
Title: A Comparative Evaluation of Subgingivally Delivered Chlorhexidine, Silk Fibroin and Combination of Fibroin and Chlorhexidine as Local Drug Delivery in Periodontitis - A Randomized Control Trial
Brief Title: Local Delivery of Silk Fibroin and Chlorhexidine
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Krishnadevaraya College of Dental Sciences & Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02_D012_126027
Record Dates: First submitted 2023-09-16; First posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Periodontal Pocket
MeSH Terms: conditions — Periodontal Pocket | interventions — Fibroins; Chlorhexidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I - Silk Fibroin (Experimental): test group 1 is treated with silk fibroin
  Interventions: Biological: silk fibroin
- Group II -Chlorhexidine (Active Comparator): test group 2 is treated with chlorhexidine
  Interventions: Drug: Chlorhexidin
- Group III - Combination of Fibroin and Chlorhexidine (Experimental): test group 3 is treated with combination of silk fibroin and chlorhexidine
  Interventions: Biological: combination of silk fibroin and chlorhexidine

INTERVENTIONS:
Biological: silk fibroin — silk fibroin extracted from bombyx mori silk worm is processed in laboratory to form silk fibroin films
  Arms: Group I - Silk Fibroin
Drug: Chlorhexidin — chlorhexidine is used
  Other Names: chlorhexidine
  Arms: Group II -Chlorhexidine
Biological: combination of silk fibroin and chlorhexidine — combination of silk fibroin and chlorhexidine is used
  Arms: Group III - Combination of Fibroin and Chlorhexidine

SUMMARY:
The current study is a prospective randomised split mouth study to evaluate the effect of Silk fibroin as drug delivery system while simultaneously assessing the efficacy of silk fibroin in comparison to chlorhexidine.

DETAILED DESCRIPTION:
Fifteen healthy individuals satisfying the inclusion and exclusion criteria were recruited for the study. A detailed, thorough medical and dental history was obtained and each patient was subjected to comprehensive clinical and radiological examination. All patients were informed about the nature of the study, procedure involved, potential benefits and risks associated with procedure and written informed consent were obtained from all patients.All the patients underwent scaling and root planing.

Following randomization, the site will be assigned to one of the three study groups.

1. Group I (SRP+ Silk Fibroin)
2. Group II (SRP+ Chlorhexidine)
3. Group III (SRP+ Combination of Fibroin and Chlorhexidine) Periodotal pack was placed and patient was recalled after 21days, 1 month and 3 month for the follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with age between 30-50 years.
2. Patients with stage I/ II with Grade A/ B periodontitis according to 2017 World workshop classification of periodontal disease will be considered.
3. Patients with localized periodontal pockets.
4. Patients willing to participate in the study.

Exclusion Criteria:

1. Patients with known systemic diseases.
2. Non complaint patients.
3. Patients who received any surgical or nonsurgical therapy 6 months before the start of the study.
4. Pregnant or lactating females.
5. Use of systemic antibiotics in the past 6 months.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Probing pocket Depth (PPD) | 3 months
  measured using a UNC-15 probe (university of North Carolina-15 periodontal probe- Hu-Friedy, Chicago, IL, USA
Relative attachment level (RAL) | 3 months
  measured by placing the acrylic stent on the selected teeth using UNC-15 probe (university of North Carolina-15 periodontal probe- Hu-Friedy, Chicago, IL, USA)

SECONDARY OUTCOMES:
Plaque Index | 3 months
  measured on the tooth surface using a probe
Gingival index | 3 month
  measured on the tooth surface using a probe
Modified Sulcus Bleeding Index | 3 months
  measured on the tooth surface using a probe